CLINICAL TRIAL: NCT00353509
Title: Prospective Mono-center Clinical Study to Evaluate the Safety and Effectiveness of an Intracardiac Septal Closure Device in Patients With Atrial Septum Defect (ASD)
Brief Title: Safety and Effectiveness Study of the Solysafe Septal Occluder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carag AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006.1621
Record Dates: First submitted 2006-07-16; First posted 2006-07-18 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Atrial Septal Defects
MeSH Terms: conditions — Heart Septal Defects, Atrial

INTERVENTIONS:
Device: Device Closure of a Septal Defect

SUMMARY:
Prospective mono-center clinical study to evaluate the safety and effectiveness of an intracardiac septal closure device in patients with atrial septum defect (ASD)

ELIGIBILITY:
Inclusion Criteria:

* ASD

Exclusion Criteria:

* Criteria that exclude catheterization (e.g. too small size, DIC, high risk of bleeding such as coagulation or clotting disorders)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ida Jovanovic, Prof. Dr., Principal Investigator — University Children's Hospital Belgrade
Locations (1):
- University Childen's Hospital, Belgrade, Serbia